CLINICAL TRIAL: NCT04494841
Title: Addressing Feasibility of the DuoTherm in Acute and Chronic Low Back Pain
Brief Title: Usability of a Multimodal External Neuromodulatory Device to Relieve Acute Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MMJ Labs LLC (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Sport and Spine Rehab Clinical Research Foundation (Other)
Responsible Party: Principal Investigator, Amy Lynn Baxter, Principal Investigator, MMJ Labs LLC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: UsabilityDuoTherm; 4R44DA049631 (NIH)
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Results first posted 2022-10-21 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Low Back Pain; Low Back Sprain; Low Back Pain, Recurrent
Keywords: Medical Device; Buzzy; Vibration; thermomechanical
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Consecutive low back pain patients were offered to try a new device and give feedback on a prototype. Once the feedback was obtained, the changes were incorporated into a production-ready model and re-evaluated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- DuoTherm VibraCool Back Device (Experimental): Patients will be offered a pain relief belt device incorporating multiple speeds of vibration and optional heat, cold, and pressure delivered through a sculpted metal plate. They will be able to choose from 8 patterns of vibration with the multiple motors (50, 100, 200Hz), and hot or cold, and will wear the device for 20 minutes.
  Interventions: Device: Duotherm VibraCool Back Device

INTERVENTIONS:
Device: Duotherm VibraCool Back Device — Low back plate belt with mechanicothermal and pressure intervention options.

SUMMARY:
Ten patients with acute or chronic low back pain will be invited to try a multimodal device for 20 minutes. Pain will be recorded prior to and after use, and feedback on the device will be elicited.

DETAILED DESCRIPTION:
To facilitate data collection of a short-term intervention, the investigators chose to enroll patients from a mixed physical therapy/chiropractic practice with demographic and economic diversity in the metro Washington area. The neuromodulatory device will have patient controlled frequencies at 50Hz, 100Hz, and 180Hz attached to a 12 x 22 cm metal plate ergonomically curved to fit the low back. The device will be wearable with a neoprene belt on both sides for patients to adjust pressure. The metal pocket in our device holds a 221g clay pack capable of being frozen to 15F or heated to 110F or patient tolerance, with 30 minute thermal capacity. A convenience sample of 10 patients at the clinic was invited to give feedback on the prototype device after informed consent. Changes suggested were incorporated and after informed consent a second group of ten gave will give feedback with the production-ready device.

ELIGIBILITY:
Inclusion Criteria:

* Acute or chronic low back pain as chief complaint
* Capacity to understand all relevant risks and potential benefits of the study (informed consent);
* Willingness to communicate information

Exclusion Criteria:

* Radicular pain likely reflecting a surgical or mechanical problem
* BMI greater than 30 (device won't fit)
* Sensitivity to cold or vibration (e.g Raynaud's or Sickle Cell Disease)
* Diabetic neuropathy rendering a patient unable to determine if the device is too hot
* New neurologic deficits
* Skin lesions over the low back area
* Contraindication to any medication for pain management that would impact analgesic use record
* Inability to apply DuoTherm

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Yes based on self-representation
Enrollment: 20 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Baxter, MD, Principal Investigator — MMJ Labs LLC
Locations (1):
- Sport and Spine Rehab Clinic, Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the clinical results reported in any publications, after deidentification, will be available for a period of 36 months after publication to achieve approved aims of any researcher who provides a methodologically sound proposal. Proposals should be directed to info@mmjlabs.com. To gain acccess, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, CSR
Time Frame: 36 months after publication
Access Criteria: researchers providing approved methodologically sound proposals

REFERENCES:
- [Background] Stumbo SP, Yarborough BJ, McCarty D, Weisner C, Green CA. Patient-reported pathways to opioid use disorders and pain-related barriers to treatment engagement. J Subst Abuse Treat. 2017 Feb;73:47-54. doi: 10.1016/j.jsat.2016.11.003. Epub 2016 Nov 15. PMID 28017184
- [Background] Darnall BD, Colloca L. Optimizing Placebo and Minimizing Nocebo to Reduce Pain, Catastrophizing, and Opioid Use: A Review of the Science and an Evidence-Informed Clinical Toolkit. Int Rev Neurobiol. 2018;139:129-157. doi: 10.1016/bs.irn.2018.07.022. Epub 2018 Aug 6. PMID 30146045
- [Background] Davis CS, Lieberman AJ, Hernandez-Delgado H, Suba C. Laws limiting the prescribing or dispensing of opioids for acute pain in the United States: A national systematic legal review. Drug Alcohol Depend. 2019 Jan 1;194:166-172. doi: 10.1016/j.drugalcdep.2018.09.022. Epub 2018 Nov 3. PMID 30445274
- [Background] Ballard A, Khadra C, Adler S, Trottier ED, Le May S. Efficacy of the Buzzy Device for Pain Management During Needle-related Procedures: A Systematic Review and Meta-Analysis. Clin J Pain. 2019 Jun;35(6):532-543. doi: 10.1097/AJP.0000000000000690. PMID 30829735
- [Background] Lurie RC, Cimino SR, Gregory DE, Brown SHM. The effect of short duration low back vibration on pain developed during prolonged standing. Appl Ergon. 2018 Feb;67:246-251. doi: 10.1016/j.apergo.2017.10.007. Epub 2017 Nov 1. PMID 29122196
- [Background] Ueki S, Yamagami Y, Makimoto K. Effectiveness of vibratory stimulation on needle-related procedural pain in children: a systematic review. JBI Database System Rev Implement Rep. 2019 Jul;17(7):1428-1463. doi: 10.11124/JBISRIR-2017-003890. PMID 31021972
- [Derived] Baxter AL, Thrasher A, Etnoyer-Slaski JL, Cohen LL. Multimodal mechanical stimulation reduces acute and chronic low back pain: Pilot data from a HEAL phase 1 study. Front Pain Res (Lausanne). 2023 Apr 26;4:1114633. doi: 10.3389/fpain.2023.1114633. eCollection 2023. PMID 37179530

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DuoTherm VibraCool Back Device
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | DuoTherm VibraCool Back Device
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.9 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 18
  White | 1
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain: Visual Analog Scale (VAS)
Description: Difference in 10 cm VAS printed on paper from 0 (no pain) to 10 (most pain) before and after use of the device, higher value indicates a greater pain reduction, 1.8 cm is considered clinically relevant.
Time Frame: Before use of device (baseline) and after use of device approximately 30 minutes - 20 minutes of use, with 10 minutes for evaluation
Measure: Mean (Standard Deviation); unit: units on a scale (centimeters)
Arm/Group | DuoTherm VibraCool Back Device
Number analyzed (Participants) | 20
units on a scale (centimeters) | 2.1 (1.4)

2. Primary Outcome: Participants' Choice in Thermal Options
Description: One of four options: hot, cold, none, both
Time Frame: 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | DuoTherm VibraCool Back Device
Number analyzed (Participants) | 20
Participants
  Hot | 9
  Cold | 11
  None | 0
  Both | 0

3. Primary Outcome: Would You Recommend
Description: Binary approval or disapproval of device
Time Frame: After 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | DuoTherm VibraCool Back Device
Number analyzed (Participants) | 20
Participants
  Approve | 20
  Disapprove | 0

4. Secondary Outcome: Subjective Pain Relief
Description: 7-item Likert scale of 1 (much worse) to 7 (much better) pain relief over the time of the study
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DuoTherm VibraCool Back Device
Number analyzed (Participants) | 20
score on a scale | 5.3 (0.98)

ADVERSE EVENTS:
Time Frame: 4 hours
Description: 20 patients will be evaluated for adverse events, mortality, or other not serious adverse events.
Arm/Group | DuoTherm VibraCool Back Device
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/41/NCT04494841/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/41/NCT04494841/ICF_001.pdf